CLINICAL TRIAL: NCT05835856
Title: e-VITA: European-Japanese Virtual Coach for Smart Ageing (WAVE II)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: INRCA_005_2023
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Older Adults; Quality of Life
Keywords: virtual coach; older adults; technological system; quality of life; usability; well-being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- NAO robot group (Experimental)
  Interventions: Device: Virtual coach with NAO robot
- Google Nest Hub (2e generation) group (Experimental)
  Interventions: Device: Virtual coach with Google Nest Hub (2e generation) group
- Gatebox group (Experimental)
  Interventions: Device: Virtual coach with Gatebox device
- CelesTE robot group (Experimental)
  Interventions: Device: virtual coach with CelesTE robot
- Control group (Other)
  Interventions: Other: booklet

INTERVENTIONS:
Device: Virtual coach with NAO robot — The coaching device used is the softbank NAO 5 and NAO 6 humanoid interactive mobile robot. These robot platform allows multimodal natural language interaction and robot autonomous movement.
  Arms: NAO robot group
Device: Virtual coach with Google Nest Hub (2e generation) group — The coaching device used is Google Nest Hub (2e generation). This is a connected speaker enriched with a 7-chip touch screen. It has a loudspeaker and 3 microphones, making interaction possible.
  Arms: Google Nest Hub (2e generation) group
Device: Virtual coach with Gatebox device — The coaching device used is the Gatebox, a hologram like device which the user can interact. There are internal sensors such as a camera and a microphone allow the user to converse with the projected character. It connects to the Internet via a wireless LAN. With infrared rays and Bluetooth, it can also be connected to household appliances and other devices.
  Arms: Gatebox group
Device: virtual coach with CelesTE robot — The coaching device used is the CelesTE robot, a prayer companion designed for Christian Catholic users.The intended main function of CelesTE is to be a "guardian angel", especially thought for elderly people. It can be a prayer companion, and contains a vast number of teachings, including the whole Bible. Its AI is capable of keeping a short conversation, in which the user may ask and receive an answer about a sensitive topic (such as happiness, death, faith, etc.). It can also printout a selection of contents.
  The coaching device CelesTE will be substituted by DarumaTO for the Japanese centers.
  Arms: CelesTE robot group
Other: booklet — Participant in the control group will receive a booklet containing information and activities on well-being
  Arms: Control group

SUMMARY:
The study is a multicentre Proof-of-Concept. The general objective of the e-VITA project is to develop a personalized virtual coach capable of interacting with its elderly interlocutor. The experimentation will be carried out in 4 sites: Italy, France, Germany and Japan.

DETAILED DESCRIPTION:
The general objective of the e-VITA project is to improve well-being for older adults and thereby promote active and healthy ageing, contribute to independent living, and reduce risks of social exclusion of older adults by making use a virtual coach by 240 healthy older adults recruited from Europe (France, Germany and Italy) and Japan. The study is a multicenter Proof-of-Concept study with a duration of the intervention of six months.

The multidisciplinary consortium collaborating in this project will develop an innovative ICT-based virtual coaching system to detect subtle changes in physical, cognitive, psychological and social domains of older adult's daily life. The e-VITA virtual coach will thus provide personalized recommendations and interventions, for sustainable wellbeing in a smart living environment at home.

The different components of the system are:

* Coaches, consisting of social robots, that will interact with the users and are guided by apps;
* Sensors (both wearable and domestic) to detect physiological parameters, physical activities, and behavior of the users; these sensors are: the Huawei smart band (wearable), the NeU device (wearable), and the DeltaDore system (domestic).
* Smartphones (the chatbot to provide insights, suggestion, and stimulation about healthy nutrition and physical exercise; the social platform to encourage users to share their interests).

These components (coaches, sensors, chatbot and social platform) together with a main software named Use Cases Configurator (UCC) constitute the Virtual Coach.

ELIGIBILITY:
Inclusion Criteria:

* Able to stand and walk unaided;
* No acute or untreated medical problems;
* Montreal Cognitive Assessement test (MOCA) ≥ 22;
* Geriatric Depression Scale (GDS) < 9;
* Short performance physical battery (SPPB) ≥ 7
* Clinical Frailty Scale score between 2 and 4.

Exclusion Criteria:

* Use of active implant or not-implant medical devices;
* Allergy to nichel;
* A myocardial infarction or stroke within 6 months;
* Painful arthritis, spinal stenosis, amputation, painful foot lesions or neuropathy limiting balance and mobility;
* Uncontrolled hypertension;
* Pacemaker or implantable cardioverter defibrillator;

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Quality of Life | baseline and 6 months later
  The EQ-5D-5L scale consists of five dimensions: mobility, independence, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, mild problems, moderate problems, severe problems and extreme problems. The participant is asked to indicate his/her health status by ticking the box corresponding to the most appropriate statement in each of the five dimensions. The numbers from the five dimensions can be combined into a 5-digit number that describes the health status of the participant.

SECONDARY OUTCOMES:
Change in usability | At 3 and 6 months from baseline
  The System Usability Scale (SUS) is a reliable tool for measuring usability. It consists of a10 item questionnaire with five response options for respondents from 'Strongly agree' to 'Strongly disagree'.
Change in frailty status | baseline and 6 months later
  The Clinical Frailty Scale (CFS) divides the older participants into 9 classes based on the information provided by them and their relatives: between 1 and 3 the patient is non-frail, pre-frail if 4, he is frail from 5 to 9.
Change in nutritional capacity | baseline and 6 months later
  The Short Food frequency questionnaires scale (FFQ) is used to estimate the frequency of daily food intake over a period of time. The FFQ asks for the frequency of certain food intake (once daily, once or twice a week, once or twice a month), and the approximate serving size. The questionnaire asks for information on the habitual intake of the food and is not to quantify the actual amount of nutrients ingested.
Change in affinity with technology | baseline and 6 months later
  The Affinity for Technology Interaction (ATI) measures a person's interaction-related affinity with technology. It consists of a total of nine items and uses a six-point Likert scale from 1 = completely disagree to 6 = completely agree.
Change in cognitive status | baseline and 6 months later
  Montreal Cognitive Assessment (MoCA) is a cognitive test validated as a highly sensitive tool for early detection of mild cognitive impairment (MCI). Scores on the MoCA range from zero to 30. A score of 26 and higher is considered normal.
Change in psychological mood | baseline and 6 months later
  The Geriatric Depression scale 5-items version (GDS-5 items) questionnaire assesses the current condition of the patient's mood. Scores >1 are indicative for depression.
Change in performance status | baseline and 6 months later
  Short Physical Performance Battery (SPPB) is a short battery of tests designed to assess the function of the lower limbs. This scale consists of 3 different sections: balance assessment, evaluation of walking on 4 linear meters, evaluation of the ability to perform, for 5 consecutive times, the sit to stand from a chair, without using the upper limbs. The total scale score therefore has a range from 0 to 12. A total score below 10 indicates frailty and a high risk of disability and falls.
Change in person's need for technology | baseline and 6 months later
  The Assistive Technology Device Predisposition Assessment (ATDPA-5 - scales B and E) assesses the person's need for technology. It has two parts. A part on the individual with 9 items assessing functional capacities and 11 items on well-being. These first 20 items are to be filled in on a Likert scale of 5, ranging from 1: poor/not satisfied to 5: excellent/very satisfied. Finally, this last part also assesses personal and psychosocial characteristics. There is no threshold value for these last items. The second part deals with technological tools with 12 items highlighting their expectations in terms of benefits towards three technological tools. There is no threshold for this scale, but the scores range from 0 to 60 (sum of the statements).

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Bevilacqua, Study Director — IRCCS INRCA, Ancona, Italy
Locations (4):
- Broca Hospital, Paris, France
- Diocesan Caritas Association for the Archdiocese of Cologne, Cologne, Germany
- IRCCS INRCA Hospital, Ancona, Italy
- Tohoku University -Smart Ageing Research Center, Miyagi, Japan